CLINICAL TRIAL: NCT06284447
Title: Barriers to Cervical Cancer Screening
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-004500; NCI-2024-00181 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-004500 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Participants complete a survey on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non interventional study

SUMMARY:
This study evaluates barriers to cervical cancer screening among non-compliant women.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To further identify barriers to cervical cancer screening in women, we will identify non-compliant patients and survey them to better understand barriers that have led to inadequate screening.

OUTLINE: This is an observational study.

Participants complete a survey on study.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 21-65
* Non-compliant for cervical cancer screening within Mayo Clinic Primary Care

Exclusion Criteria:

* Women less than 21 or older than 65
* Complaint for cervical cancer screening within Mayo Clinic Primary Care
* Women who decline participation

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 21-65 that are non-compliant for cervical cancer screening within the Mayo Clinic Health System
Sampling Method: Non-Probability Sample
Enrollment: 2216 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Identify barriers to cervical cancer screening | Baseline
  Participants will receive a brief "Pap Smear Barriers Survey" (likely completed in 5-15 minutes) which asks yes/no/no preference questions regarding potential barriers to cervical cancer screening. Responses will be compared regionally and by Mayo Clinic Health System site.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany A. Strelow, DSMc, PA-C, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials